CLINICAL TRIAL: NCT04114526
Title: Collaboration to Develop and Pilot Test a Community Health Advisor Smoking Cessation Program for Durham Public Housing Residents
Brief Title: Durham Housing Authority (DHA) Community Health Advisor (CHA) Smoking Cessation Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00100099
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Health Advisor 4-step Program (Experimental)
  Interventions: Other: Nicotine Replacement Therapy

INTERVENTIONS:
Other: Nicotine Replacement Therapy — CHAs meet with all interested residents to discuss taking steps towards quitting. The CHAs follow a four step program with all participant 1) get to know the resident and their smoking, 2) Assess what the resident is ready to do to take steps towards quitting, 3) discuss using nicotine replacement therapy (NRT) in the form of patches, gum or lozenges, 4) set one goal for taking steps towards quitting. CHAs will attempt to follow up with participants after the initial encounter. There is no limit on the number of times the CHA may talk with the participants. Some follow interactions will be brief encounters in the neighborhood, while others will be at scheduled. All contacts with each participant will be tracked.
  We will provide up to 6 weeks of NRT patches, gum and lozenges to participants who are interested in using NRT to help them quit.

SUMMARY:
Recent policy from the U.S. Department of Housing and Urban Development (HUD) mandates that all public housing units go smoke-free by August 2018. Residents in public housing units have little access to proven cessation interventions and support is imperative to increase quitting success and is currently lacking in these communities;' thus this mandate is causing stress without providing resources to quit. Using a Community Engaged Research (CEnR) approach, we propose to partner the Durham County Department of Public Health and the Durham Housing Authority to develop sustainable Community Health Advisor tobacco cessation program that can be implemented in public housing communities. To achieve this goal, we plan to build on our previous collaborations to 1) form a team of previously identified DHA residents who are activated to support smoking cessation among public housing residents who can serve as Community Health Advisors and deliver cessation interventions in DHA properties, and 2) co-develop and pilot test a Community Health Advisor smoking cessation program to promote linkages with cessation services and to provide cessation education to DHA residents. This collaboration builds on our previous work to understand barriers and identify solutions for supporting smoking cessation among DHA residents. We will work with Community Health Advisors to develop an intervention and conduct a pilot study with up to 30 participants, Our primary outcomes are feasibility and acceptability of the co-development cessation intervention. We will collect survey data for the pilot in REDCap. Potential risks of study participation include breach of confidentiality with regard to identifiable personal information and questions that might make participants feel uncomfortable.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* current smoker (smoked in the last seven days)
* planning on quitting in the next 6 months
* speak English
* currently living in DHA property

Exclusion Criteria:

* less than18 years of
* cognitive impairment
* planning to move from the property in the next 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Number of people who enroll in the study as measured by enrollment log. | 4 months
Number of people that interact with community health advisors | 5 months
Number of participants who rate the intervention as helpful for quitting based on survey questionnaire. | 5 months
Change in number of cigarettes smoked per day as measured by questionnaire | Baseline and day 28
Change in smoking cessation motivation will be self-reported on a 7-point scale. | Baseline and day 28
  1=not at all motivated and 7=completely motivated.
Change in smoking status as measured by self-reports. | Baseline and day 28
  Participants will be asked on a questionnaire, "Have you smoked in the last 7 days even a puff" and will have the option of answering "yes" or "no".
Frequency of interaction with community health advisors during intervention period will be calculated from self-reports. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Fish, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcomes will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.